CLINICAL TRIAL: NCT03166150
Title: Urinary Incontinence, Mobility & Muscle Function in Older Women: Functional Assessment and Muscle Evaluation Through Exercise (FAME) Trial
Brief Title: Functional Assessment and Muscle Evaluation Through Exercise Trial
Acronym: FAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Collaborators: National Hispanic Council on Aging (NHCOA) (Other)
Responsible Party: Principal Investigator, Tatiana Sanses, MD FACOG FPMRS, Associate Professor, Chief, Female Pelvic Medicine & Reconstructive Surgery, Urogynecology, Howard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-MED-21
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2020-09

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Pelvic Floor Disorder; Pelvic Floor Muscle; Strength; Disability; Aging; Atrophy; Exercise; Magnetic Resonance Imaging; Fatty Infiltration; Physical Therapy; Multi-modal Rehabilitation; Stress Urinary Incontinence; Urge Urinary Incontinence; Mixed Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders; Atrophy; Motor Activity; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-modal rehabilitation program (Experimental): 12 weeks of various exercises
  Interventions: Other: Multi-modal rehabilitation program
- Pelvic Floor Physical therapy (Active Comparator): 12 weeks of standard pelvic floor physical therapy
  Interventions: Other: Pelvic Floor Physical therapy

INTERVENTIONS:
Other: Multi-modal rehabilitation program — Patients will receive 12 weeks of exercises.
  Arms: Multi-modal rehabilitation program
Other: Pelvic Floor Physical therapy — Pelvic Floor Physical therapy
  Arms: Pelvic Floor Physical therapy

SUMMARY:
The purpose of this study is to decrease rates of urinary incontinence in older women by building strength in the pelvic and lower body muscle through exercise and rehabilitation.

DETAILED DESCRIPTION:
This study will provide data on benefits of combination the multimodal strengthening and aerobic conditioning rehabilitation program with pelvic floor muscle training and will help to characterize changes in pelvic floor and lower extremity muscles in older women with urinary incontinence.

The study focuses on a patient-centered approach to improve overall physical function in older women. The study will evaluate the incremental benefit of endurance and lower extremity muscle strengthening in addition to benefits from pelvic floor muscle training. We anticipate that this approach will decrease rates of urinary incontinence because the proposed intervention will focus on prevention of functional decline through endurance, strength, and balance training among older women.

The study will evaluate the pathophysiology of urinary incontinence in older women through evaluation of pelvic floor and lower extremities muscles with an innovative MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 65 years older
2. Symptomatic UI
3. Symptoms ≥ 3 months
4. Episodes of UI on 3-day bladder diary
5. Stress, urgency, and mixed UI

Exclusion Criteria:

1. Women unable to have functional assessment and/or complete bladder diary
2. Impaired mental status (MMSE <25)
3. Post-void residual ≥ 150 ml
4. Non-ambulatory (wheelchair bound), unable to complete mobility assessments
5. Hematuria
6. Urinary tract infection
7. Continuous Incontinence
8. Pelvic Organ prolapse > stage 2
9. Fecal impaction (no BM within 1 week), severe congestive heart failure (leg swelling edema 2+), uncontrolled diabetes (positive urine glucose Dipstick test)
10. Women with significant neurological or musculoskeletal conditions that compromise mobility (stroke, multiple sclerosis, amyotrophic atrophic lateral sclerosis, severe rheumatoid arthritis)
11. Women with contraindications to undergo MRI including claustrophobia.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Reduction of UI episodes | 12 weeks
  The primary outcome of this study is reduction in urinary incontinence episodes after multi-modal rehabilitation program compared to standard pelvic floor physical therapy.

SECONDARY OUTCOMES:
muscle strength | 12 weeks
  functional assessment
muscle quality | 12 weeks
  MRI evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Sanses, M.D., Principal Investigator — Howard University
Locations (1):
- Howard University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunskaar S, Arnold EP, Burgio K, Diokno AC, Herzog AR, Mallett VT. Epidemiology and natural history of urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2000;11(5):301-19. doi: 10.1007/s001920070021. PMID 11052566
- [Background] Huang AJ, Brown JS, Thom DH, Fink HA, Yaffe K; Study of Osteoporotic Fractures Research Group. Urinary incontinence in older community-dwelling women: the role of cognitive and physical function decline. Obstet Gynecol. 2007 Apr;109(4):909-16. doi: 10.1097/01.AOG.0000258277.01497.4b. PMID 17400853
- [Background] Hirsch JF, Rose CS, Pierre-Kahn A, Renier D, Hoppe-Hirsch E. Neurosurgery with craniotomy and CT stereotactic guidance in the treatment of intracerebral space-occupying lesions. Childs Nerv Syst. 1990 Sep;6(6):323-6. doi: 10.1007/BF00298277. PMID 2257544
- [Background] Harris SS, Link CL, Tennstedt SL, Kusek JW, McKinlay JB. Care seeking and treatment for urinary incontinence in a diverse population. J Urol. 2007 Feb;177(2):680-4. doi: 10.1016/j.juro.2006.09.045. PMID 17222656
- [Background] Hannestad YS, Rortveit G, Hunskaar S. Help-seeking and associated factors in female urinary incontinence. The Norwegian EPINCONT Study. Epidemiology of Incontinence in the County of Nord-Trondelag. Scand J Prim Health Care. 2002 Jun;20(2):102-7. PMID 12184708
- [Background] Morrill M, Lukacz ES, Lawrence JM, Nager CW, Contreras R, Luber KM. Seeking healthcare for pelvic floor disorders: a population-based study. Am J Obstet Gynecol. 2007 Jul;197(1):86.e1-6. doi: 10.1016/j.ajog.2007.02.051. PMID 17618770
- [Background] Stickley A, Santini ZI, Koyanagi A. Urinary incontinence, mental health and loneliness among community-dwelling older adults in Ireland. BMC Urol. 2017 Apr 8;17(1):29. doi: 10.1186/s12894-017-0214-6. PMID 28388898
- [Background] Yip SO, Dick MA, McPencow AM, Martin DK, Ciarleglio MM, Erekson EA. The association between urinary and fecal incontinence and social isolation in older women. Am J Obstet Gynecol. 2013 Feb;208(2):146.e1-7. doi: 10.1016/j.ajog.2012.11.010. Epub 2012 Nov 15. PMID 23159696
- [Background] Jerez-Roig J, Santos MM, Souza DL, Amaral FL, Lima KC. Prevalence of urinary incontinence and associated factors in nursing home residents. Neurourol Urodyn. 2016 Jan;35(1):102-7. doi: 10.1002/nau.22675. Epub 2014 Oct 12. PMID 25307780
- [Background] Ko Y, Lin SJ, Salmon JW, Bron MS. The impact of urinary incontinence on quality of life of the elderly. Am J Manag Care. 2005 Jul;11(4 Suppl):S103-11. PMID 16161383
- [Background] Thom DH, Haan MN, Van Den Eeden SK. Medically recognized urinary incontinence and risks of hospitalization, nursing home admission and mortality. Age Ageing. 1997 Sep;26(5):367-74. doi: 10.1093/ageing/26.5.367. PMID 9351481
- [Background] Goode PS, Burgio KL, Richter HE, Markland AD. Incontinence in older women. JAMA. 2010 Jun 2;303(21):2172-81. doi: 10.1001/jama.2010.749. PMID 20516418
- [Background] Roe B, Flanagan L, Jack B, Barrett J, Chung A, Shaw C, Williams K. Systematic review of the management of incontinence and promotion of continence in older people in care homes: descriptive studies with urinary incontinence as primary focus. J Adv Nurs. 2011 Feb;67(2):228-50. doi: 10.1111/j.1365-2648.2010.05481.x. Epub 2010 Nov 24. PMID 21105895
- [Background] Roe B, Flanagan L, Jack B, Shaw C, Williams K, Chung A, Barrett J. Systematic review of descriptive studies that investigated associated factors with the management of incontinence in older people in care homes. Int J Older People Nurs. 2013 Mar;8(1):29-49. doi: 10.1111/j.1748-3743.2011.00300.x. Epub 2011 Dec 19. PMID 22182302
- [Background] Tannenbaum C, Agnew R, Benedetti A, Thomas D, van den Heuvel E. Effectiveness of continence promotion for older women via community organisations: a cluster randomised trial. BMJ Open. 2013 Dec 10;3(12):e004135. doi: 10.1136/bmjopen-2013-004135. PMID 24334159
- [Background] Willis-Gray MG, Sandoval JS, Maynor J, Bosworth HB, Siddiqui NY. Barriers to urinary incontinence care seeking in White, Black, and Latina women. Female Pelvic Med Reconstr Surg. 2015 Mar-Apr;21(2):83-6. doi: 10.1097/SPV.0000000000000100. PMID 25185610
- [Background] MacLachlan LS, Rovner ES. New treatments for incontinence. Adv Chronic Kidney Dis. 2015 Jul;22(4):279-88. doi: 10.1053/j.ackd.2015.03.003. PMID 26088072
- [Background] Adelmann PK. Prevalence and detection of urinary incontinence among older Medicaid recipients. J Health Care Poor Underserved. 2004 Feb;15(1):99-112. doi: 10.1353/hpu.2004.0001. PMID 15359977
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Vaughan CP, Goode PS, Burgio KL, Markland AD. Urinary incontinence in older adults. Mt Sinai J Med. 2011 Jul-Aug;78(4):558-70. doi: 10.1002/msj.20276. PMID 21748744
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Coyne KS, Wein A, Nicholson S, Kvasz M, Chen CI, Milsom I. Economic burden of urgency urinary incontinence in the United States: a systematic review. J Manag Care Pharm. 2014 Feb;20(2):130-40. doi: 10.18553/jmcp.2014.20.2.130. PMID 24456314
- [Background] Paiva LL, Ferla L, Darski C, Catarino BM, Ramos JG. Pelvic floor muscle training in groups versus individual or home treatment of women with urinary incontinence: systematic review and meta-analysis. Int Urogynecol J. 2017 Mar;28(3):351-359. doi: 10.1007/s00192-016-3133-2. Epub 2016 Sep 9. PMID 27613622
- [Background] Waddie B, Meawad E.
- [Background] Leroy LS, Lopes MH, Shimo AK. Urinary incontinence in women and racial aspects: a literature review. Text Contex Nursing, 2012 Jul-Sept; 21(3):692-701
- [Background] Lammers K, Kluivers KB, Vierhout ME, Prokop M, Futterer JJ. Inter- and intraobserver reliability for diagnosing levator ani changes on magnetic resonance imaging. Ultrasound Obstet Gynecol. 2013 Sep;42(3):347-52. doi: 10.1002/uog.12462. PMID 23494887
- [Background] Morgan DM, Umek W, Stein T, Hsu Y, Guire K, DeLancey JO. Interrater reliability of assessing levator ani muscle defects with magnetic resonance images. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Jul;18(7):773-8. doi: 10.1007/s00192-006-0224-5. Epub 2006 Oct 17. PMID 17043740
- [Background] Visser M, Goodpaster BH, Kritchevsky SB, Newman AB, Nevitt M, Rubin SM, Simonsick EM, Harris TB. Muscle mass, muscle strength, and muscle fat infiltration as predictors of incident mobility limitations in well-functioning older persons. J Gerontol A Biol Sci Med Sci. 2005 Mar;60(3):324-33. doi: 10.1093/gerona/60.3.324. PMID 15860469
- [Background] Addison O, Young P, Inacio M, Bair WN, Prettyman MG, Beamer BA, Ryan AS, Rogers MW. Hip but not thigh intramuscular adipose tissue is associated with poor balance and increased temporal gait variability in older adults. Curr Aging Sci. 2014;7(2):137-43. doi: 10.2174/1874609807666140706150924. PMID 24998419
- [Background] Inacio M, Ryan AS, Bair WN, Prettyman M, Beamer BA, Rogers MW. Gluteal muscle composition differentiates fallers from non-fallers in community dwelling older adults. BMC Geriatr. 2014 Mar 25;14:37. doi: 10.1186/1471-2318-14-37. PMID 24666603
- [Background] Kiyoshige Y, Watanabe E. Fatty degeneration of gluteus minimus muscle as a predictor of falls. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):59-61. doi: 10.1016/j.archger.2014.07.013. Epub 2014 Aug 1. PMID 25440137
- [Background] Bogunovic L, Lee SX, Haro MS, Frank JM, Mather RC 3rd, Bush-Joseph CA, Nho SJ. Application of the Goutallier/Fuchs Rotator Cuff Classification to the Evaluation of Hip Abductor Tendon Tears and the Clinical Correlation With Outcome After Repair. Arthroscopy. 2015 Nov;31(11):2145-51. doi: 10.1016/j.arthro.2015.04.101. Epub 2015 Jul 15. PMID 26188781
- [Background] Robert B. Wallace ARH. Documentation of Physical Functioning Measured in the Health and Retirement Study and the Asset and Health Dynamics among the Oldest Old Study. 2004.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] American College of Sports Medicine, Thompson WR, Gordon NF, Pescatello LS. ACSM's guidelines for exercise testing and prescription. Philadelphia: Wolters Kluwer/Lippincott Williams & Wilkins; 2010.
- [Background] American College of Sports Medicine, Ehrman JK, De-Jong A, Sanderson B, Swain D, Swank A, Womack C. ACSM's Resource Manual for Guidelines for Exercise Testing and Prescription. Seventh edition. Philadelphia: LWW; 2013. 896 p.
- [Background] Hay-Smith J, Herderschee R, Dumoulin C, Herbison P. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women: an abridged Cochrane systematic review. Eur J Phys Rehabil Med. 2012 Dec;48(4):689-705. PMID 23183454
- [Background] Felicissimo MF, Carneiro MM, Saleme CS, Pinto RZ, da Fonseca AM, da Silva-Filho AL. Intensive supervised versus unsupervised pelvic floor muscle training for the treatment of stress urinary incontinence: a randomized comparative trial. Int Urogynecol J. 2010 Jul;21(7):835-40. doi: 10.1007/s00192-010-1125-1. Epub 2010 Feb 24. PMID 20179901
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Pearson S, Temple L, Bishop T, Ukaegbu A, Alden J, Kwagyan J, Sanses TVD. Community-based Versus Traditional Research Among Older Minority Women With Urinary Incontinence. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):201-206. doi: 10.1097/SPV.0000000000001089. Epub 2021 Aug 11. PMID 34387261